CLINICAL TRIAL: NCT04416724
Title: Canadian Pseudoexfoliation Glaucoma Trial: Comparison of Phacoemulsification Versus Selective Laser Trabeculoplasty as Initial Treatment for Pseudoexfoliation Glaucoma
Brief Title: Phacoemulsification vs SLT as Initial Treatment for Pseudoexfoliation Glaucoma
Acronym: CANPEX1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Glaucoma Research Society of Canada (Other); Canadian Glaucoma Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CANPEX1
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pseudoexfoliation Glaucoma
MeSH Terms: conditions — Exfoliation Syndrome | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phacoemulsification (Experimental): Main study intervention will be Phacoemulsification
  Interventions: Procedure: Phacoemulsification
- SLT (Experimental): Main study intervention will be Selective Laser Trabeculoplasty
  Interventions: Device: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Phacoemulsification — Lens removal by Phacoemulsification
  Arms: Phacoemulsification
Device: Selective Laser Trabeculoplasty — Laser application in trabecular meshwork
  Arms: SLT

SUMMARY:
The Canadian Pseudoexfoliation Glaucoma Study 1 is a randomized clinical trial that aims to compare two initial treatment options - Selective Laser Trabeculoplasty (SLT) and Phacoemulsification (PHACO) - in newly diagnosed patients with pseudoexfoliation and need to lower the intraocular pressure. Patients with pseudoexfoliation and a recent decision to lower the intraocular pressure, who also have early asymptomatic lens opacification will be recruited and randomized to receive either SLT or PHACO. Patients will be followed for 2 years according to a target IOP protocol based on the Canadian Ophthalmological Society Glaucoma guidelines. Patients who do not achieve the target IOP with the initial randomization procedure will receive IOP lowering medications. The main outcome of interest will be the proportion of subjects who need IOP lowering medications after 2 years. Secondary outcomes include IOP reduction, time to need medications, patient reported outcomes in terms of visual function, and occurrence of adverse effects. To obtain longer follow-up information beyond two years, a chart review will be done 5 and 10 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Pseudoexfoliation syndrome, detected at slit-lamp examination by exfoliative material on anterior capsule, pupil, or anterior chamber angle
2. Clinical decision to lower the IOP, as assessed by the investigator who is treating the subject, based on the presence of PXG or with IOP elevated enough to warrant treatment, even without clear evidence of optic nerve damage or visual field defect
3. Presence of asymptomatic early cataract

Exclusion Criteria:

1. Age less than 50 years old
2. Anterior chamber angle closure at gonioscopy, defined as pigmented trabeculum visible in less than 180º
3. Previous IOP lowering procedure such as trabeculoplasty, trabeculectomy, or minimally invasive glaucoma surgery
4. Previous use of IOP lowering medication for more than 6 months
5. Presence of ocular or systemic pathology or medication that could significantly influence the IOP, such as: uveitis, neovascular or traumatic glaucoma, corneal pathology influencing tonometry, use of oral steroids
6. IOP at baseline visit higher than 36 mmHg
7. Visual field damage at baseline visit with mean deviation worse than -15 dB
8. Not able or willing to provide voluntary, informed consent to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Medication-free intraocular pressure control | 2 years
  Proportion of subjects without use of intraocular pressure lowering medications

SECONDARY OUTCOMES:
Medication-free intraocular pressure control | 10 years
  Proportion of subjects without use of intraocular pressure lowering medications
Intraocular pressure change from baseline | 10 years
Number of intraocular pressure lowering medications | 10 years
Time to introduction of intraocular pressure lowering medications | 10 years
Number of adverse effects | 10 years
Score at the Glaucoma Quality of Life - 15 | 10 years
  The questionnaire GQL-15 was described in PMID: 12671469. The minimum value is 15 and the maximum is 75, with lower values indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada